CLINICAL TRIAL: NCT00006130
Title: Randomized Study of Decompression Coring Versus Conservative Therapy in Patients With Avascular Necrosis of the Hip Related to Sickle Cell Disease
Brief Title: Decompression Coring Versus Conservative Therapy in Patients With Avascular Necrosis of the Hip Related to Sickle Cell Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: NCRR-M01RR01271-5715; UNCCH-GCRC-1375
Record Dates: First submitted 2000-08-03; First posted 2000-08-04 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Bone Avascular Necrosis; Sickle Cell Anemia
Keywords: arthritis & connective tissue diseases; avascular necrosis; disease-related problem/condition; genetic diseases and dysmorphic syndromes; hematologic disorders; pain; rare disease; sickle cell anemia
MeSH Terms: conditions — Osteonecrosis; Anemia, Sickle Cell; Arthritis; Connective Tissue Diseases; Genetic Diseases, Inborn; Hematologic Diseases; Pain; Rare Diseases

INTERVENTIONS:
Procedure: Core decompression

SUMMARY:
OBJECTIVES: I. Phase II trial to determine surgical morbidity of decompression coring, including any adverse events in the perioperative period and the rate of secondary medical or surgical interventions.

II. Collect preliminary data to determine if decompression coring results in a substantial improvement in pain and mobility compared to conservative therapy in patients with avascular necrosis of the hip related to sickle cell disease.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, multicenter study. Patients are stratified according to stage of avascular necrosis (I vs II vs III). Patients are randomized into one of two treatment arms.

Arm I: Patients undergo a core biopsy and decompression of the hip followed by a standardized program of touch down or nonweight bearing with appropriate equipment and regular physical therapy for 6 weeks and then full weight bearing if tolerated.

Arm II: Patients undergo the standardized ambulation and physical therapy program as in arm I. They do not undergo any surgical procedure.

For 1 week prior to the beginning of the standardized program and during the 6 weeks of touch down or nonweight bearing, all patients complete a weekly pain and medication diary.

Patients are followed at 3 months and 6 months, then every 6 months for 1.5 years, and then annually for up to 5 years.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of stage I, II, or III avascular necrosis (AVN) by MRI or plain film imaging that is related to sickle cell disease
* Clinically moderate to severe pain originating from the hip and/or limitation of movement of the affected hip
* AVN in the contralateral hip allowed, regardless of stage, if the primary hip is eligible If both hips eligible, most symptomatic hip enrolled

Exclusion criteria:

* Non-sickle cell arthropathies
* Concurrent chronic steroids
* Chronic transfusion therapy
* Alcoholism

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 1999-06

CONTACTS AND LOCATIONS:
Overall Officials: Elliott P. Vichinsky, Study Chair — UCSF Benioff Children's Hospital Oakland
Locations (2):
- United States (2):
  - Children's Hospital of Oakland, Oakland, California
  - University of North Carolina School of Medicine, Chapel Hill, North Carolina